CLINICAL TRIAL: NCT02530736
Title: Responsiveness of the 4 Metre Gait Speed in Patients With Idiopathic Pulmonary Fibrosis and Determination of the Minimum Important Difference
Brief Title: Responsiveness and MID of 4 Metre Gait Speed in Idiopathic Pulmonary Fibrosis
Acronym: IPFRESP
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 14/LO/2247
Record Dates: First submitted 2015-05-01; First posted 2015-08-21 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Gait speed; Pulmonary Rehabilitation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IPF_RESP: Pulmonary Rehabilitation: a 6 - 8 week exercise and education programme (this is part of usual care)
  Interventions: Other: 4 metre gait speed

INTERVENTIONS:
Other: 4 metre gait speed — Measurement of usual walking speed over 4 metres. Change in walking speed is measured at baseline (pre-pulmonary rehabilitation assessment) and 8 weeks later (post-pulmonary rehabilitation assessment)
  Other Names: 4MGS

SUMMARY:
This study measures the 4 metre gait speed (4MGS) test in patients with Idiopathic Pulmonary Fibrosis (IPF). The investigators are interested to see whether usual walking speed in IPF patients changes following pulmonary rehabilitation and if it changes, what is the smallest change that is meaningful to patients.

DETAILED DESCRIPTION:
This observational study is investigating a simple test of usual walking speed, measured using the 4 metre gait speed (4MGS) test in patients with a lung disease called Idiopathic Pulmonary Fibrosis (IPF). Drug development for this disease is slow in part because there is a lack of reliable measurements that can assess effectiveness of treatment. Slow walking speed has been shown to relate to poor outcomes in older adults and people with another lung disease called Chronic Obstructive Pulmonary Disease (COPD). The investigators are interested to see whether usual walking speed in IPF patients changes following a treatment called pulmonary rehabilitation (an exercise and education programme for patients with lung disease) and if it changes, what is the smallest change that is meaningful to patients (the minimum important difference - MID). The investigators are also investigating whether the change in walking speed can predict survival, number of hospital admissions and lung disease progression. This will help inform us of the potential use of 4MGS as an outcome measure. To do this, participants who consent to taking part in the study will be timed walking at their usual walking speed over a distance of 4 metres (13.12 feet) before and after a course of pulmonary rehabilitation and follow-up 1 year after completing pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Idiopathic Pulmonary Fibrosis according to NICE guidelines referred for Pulmonary Rehabilitation
* Provided informed consent

Exclusion Criteria:

* Significant co-morbidities that would limit walking ability, exercise capacity or make exercise unsafe (e.g. unstable ischaemic heart disease, neuromuscular disease, severe hip/lower limb joint pain, peripheral vascular disease, lower limb amputation)
* Any patient whom the chief investigator feels it is unsafe to exercise (e.g. unstable cardiovascular disease)
* Any condition that precludes providing informed consent e.g. cognitive impairment or poor English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Idiopathic Pulmonary Fibrosis according to NICE guideliness referred for Pulmonary Rehabilitation
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10-17 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Change in usual walking speed measured using the 4 metre gait speed test | Change from baseline to 8 weeks
  A measure of usual walking speed

CONTACTS AND LOCATIONS:
Overall Officials: William DC Man, MD, PhD, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, Harefield, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nolan CM, Delogu V, Maddocks M, Patel S, Barker RE, Jones SE, Kon SSC, Maher TM, Cullinan P, Man WD. Validity, responsiveness and minimum clinically important difference of the incremental shuttle walk in idiopathic pulmonary fibrosis: a prospective study. Thorax. 2017 Sep 7:thoraxjnl-2017-210589. doi: 10.1136/thoraxjnl-2017-210589. Online ahead of print. PMID 28883090